CLINICAL TRIAL: NCT00526331
Title: Randomized Evaluation of Arterial Pressure Based Cardiac Output for Goal-Directed Perioperative Therapy
Brief Title: Evaluation of Arterial Pressure Based Cardiac Output for Goal-Directed Perioperative Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-0231
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2011-12

CONDITIONS: Esophageal Diseases; Gastrointestinal Diseases; Disorder of the Genitourinary System; Gynecologic Diseases; Kidney Diseases; Liver Diseases; Pancreatic Diseases; Prostate Cancer; Spinal Disease
Keywords: Perioperative Therapy; Perioperative Hydration; Arterial Pressure Based Cardiac Output; Vigileo Monitor; FloTrac Sensor; Fluid Volume; APCO
MeSH Terms: conditions — Esophageal Diseases; Gastrointestinal Diseases; Urogenital Diseases; Genital Diseases, Female; Kidney Diseases; Liver Diseases; Pancreatic Diseases; Prostatic Neoplasms; Spinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Experimental): FloTrac Sensor + Vigileo Monitor used to decide how much fluid to give during surgery.
  Interventions: Device: Vigileo Monitor; Device: FloTrac Sensor
- Control Group (Experimental): FloTrac Sensor + Vigileo Monitor only used for data collection during surgery; Standard of Care to decide fluid amount.
  Interventions: Device: Vigileo Monitor; Device: FloTrac Sensor

INTERVENTIONS:
Device: Vigileo Monitor — Study Group = The monitor and routine vital sign measurements will be used to decide how much fluid to give during surgery; Control Group = Information from the monitor will be collected and compared to the information collected from participants in Study Group.
Device: FloTrac Sensor — Device connected to the patient's arterial line and Vigileo monitor that measures fluid requirements during surgery.

SUMMARY:
The purpose of this study is to determine whether the early identification and more precise intervention of operating room (OR) patient fluid administration optimization using arterial pressure-based cardiac output (APCO) yields comparable patient outcome as fluid administration optimization using a global standard care method.

DETAILED DESCRIPTION:
THE EDWARDS VIGILEO MONITOR:

The Vigileo™ monitor measures the amount of blood the heart pumps through the body.

SCREENING TEST:

Before you can begin this study, you will have a "screening test" to help the doctor decide if you are eligible to take part in this study. Women who are able to have children must have a negative urine pregnancy test.

STUDY GROUP:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to either the Control Group or the Study Group. You will have an equal chance of being assigned to either group. You will not know to which group you have been assigned.

STUDY PARTICIPATION:

You will have a arterial catheter (small plastic tube) inserted into an artery inside your wrist at the beginning of surgery. This is used routinely (even in patients not taking part in the study) to measure your blood pressure more accurately rather than with a blood pressure cuff. It is inserted after you receive general anesthesia (numbing medicine), so you should feel no pain. If it is inserted while you are awake (based on the judgment of your anesthesiologist), then local anesthesia will be given to you to reduce discomfort.

If your doctors decide that an arterial catheter is not required as part of your routine medical care during your surgery, they will not place one for study purposes only. In that situation, you will be removed from the study, and your medical care will continue as planned by your doctors.

If the catheter is placed, the Vigileo™ monitor will be connected to the catheter and readings will be taken during the surgery. It will be disconnected at the end of surgery.

If you are in the Study Group, your doctor will use the monitor and routine vital sign measurement to decide how much fluid to give you during surgery.

If you are in the Control Group, your doctor will not know the information being collected by the monitor, as it will be collected and compared to the information collected from participants in the Study Group. The amount of fluid you received during surgery will be decided by routine vital sign measurement, as is standard of care.

ESOPHAGEAL DOPPLER:

Regardless of study group assignment, during your surgery, researchers will also connect an esophageal doppler which will also collect data on fluid volume.

The esophageal doppler is a thin, tube-like device that is placed in your throat while you are asleep. This is used routinely by doctors to assist in the administration of fluids during surgery.

The information from the doppler will be compared to the information collected from the Vigileo™ monitor. The esophageal doppler measures blood flow through your heart by ultrasound waves.

LENGTH OF STUDY:

You will be considered off study once you leave the recovery room.

FOLLOW-UP:

Researchers will be collecting information on your progress during and after surgery, including when you are allowed to leave the hospital. Your medical records will be reviewed after surgery and up to 6 months after surgery to see how you are doing and if you have had any medical problems. The kind of information researchers will be collecting is the amount of time you were in the intensive care (if any), amount of time in the hospital, any complications or problems you may have had, how well you organs are functioning, and general health information.

This is an investigational study. The Vigileo™ Monitor and esophageal doppler are FDA approved and commercially available for volume monitoring. The comparison of the monitor and doppler is investigational.

Up to 218 patients will be enrolled in this multi-center study. Up to 66 will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is in hospital for study indicated treatment.
2. Patient is able to comply with the study procedure.
3. Patient must require an indwelling radial or a femoral artery catheter.
4. Patients with an American Society of Anesthesiologists Risk Score >= 3.
5. Lee Risk Index >/= 2 (Hypertension and Pre-diabetic metabolic state).
6. Patient must be 40 kg or heavier.
7. Patient has consented to be in the trial.
8. Patient's height and weight can be accurately obtained prior to study start.
9. Patient's ability to undergo major surgery with an anticipated blood loss > 500 ml.

Exclusion Criteria:

1. Patients with contraindications for the placement of radial, femoral, or other arterial cannula.
2. Patients with contraindications for the placement of central venous cannula.
3. Patients being treated with an intra-aortic balloon pump.
4. Patients with aortic valve regurgitation.
5. Patients with atrial fibrillation.
6. Female patients with a known pregnancy confirmed by urine pregnancy test.
7. Patient is currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mena, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period of August 8, 2007 to June 30, 2008 at UT MD Anderson Cancer Center. Study recruitment done at medical clinics.
Pre-assignment Details: Study terminated by sponsor responsible for multi-center data collection and reporting. No data collection or analysis completed.
Groups:
- Overall Study: Study Group: FloTrac Sensor + Vigileo Monitor used to decide how much fluid to give during surgery; and Control Group: FloTrac Sensor + Vigileo Monitor only used for data collection during surgery while Standard of Care used to decide fluid amount.
Period: Overall Study
Arm/Group | Overall Study
Started | 55
Completed | 0
Not Completed | 55
Not completed — Sponsor Termination | 55

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 55
Age Continuous [Median (Full Range); unit: years] | 62 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay (LOS) by Participant
Description: Length of hospital stay of arterial pressure-based cardiac output (APCO) monitor participants versus the participants using the global standard care guided by esophageal Doppler, measured in days.
Time Frame: From baseline (first day of hospital stay) to release from hospital (anticipate 5 days minimally)
Population: Study terminated by sponsor without analysis due to technical reasons.
Measure: Number; unit: days
Arm/Group | Overall Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 Months
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No